CLINICAL TRIAL: NCT03555890
Title: A Single Centre, Single Dose, Open-label, Randomized, 2-part, 2-way Crossover Study to Determine the Bioequivalence of Levocetirizine Oral Disintegrating Tablet Given With Water and Without Water Compared to Levocetirizine Immediate Release Tablet in Healthy Japanese Male Subjects
Brief Title: Bioequivalence Study Between Levocetirizine Oral Disintegrating Tablet (ODT) and Levocetirizine Immediate Release Tablet (IRT)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Zensei Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 204706
Record Dates: First submitted 2018-05-09; First posted 2018-06-14 (Actual); Results first posted 2019-09-12 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Rhinitis
Keywords: Oral disintegrating tablet; Levocetirizine; Immediate release tablet; Bioequivalence; Japanese subjects
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Intervention Model Description: This study is 2-way crossover 2 part study. In Part 1, comparison of bioavailability of levocetirizine ODT and levocetirizine IRT taken with water in the fasted state will be done and In Part 2, comparison of bioavailability of levocetirizine ODT without water and levocetirizine IRT with water in the fasted state will be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Subjects of Group A: Part 1 (Experimental): Subjects in Group A will be randomized to receive levocetirizine IRT 5 mg with 150 mL water in fasted state in Period 1. After a washout period of at least 5 days, subjects will receive levocetirizine ODT 5 mg with 150 mL water in fasted state in Period 2.
  Interventions: Drug: Levocetirizine IRT 5 mg; Drug: Levocetirizine ODT 5 mg
- Subjects of Group B: Part 1 (Experimental): Subjects in Group B will be randomized to receive levocetirizine ODT 5 mg with 150 mL water in fasted state in Period 1. After a washout period of at least 5 days, subjects will receive levocetirizine IRT 5 mg with 150 mL water in fasted state in Period 2.
  Interventions: Drug: Levocetirizine IRT 5 mg; Drug: Levocetirizine ODT 5 mg
- Subjects of Group C: Part 2 (Experimental): Subjects in Group C will be randomized to receive levocetirizine IRT 5 mg with 150 mL water in fasted state in Period 1. After a washout period of at least 5 days, subjects will receive levocetirizine ODT 5 mg without water in fasted state in Period 2.
  Interventions: Drug: Levocetirizine IRT 5 mg; Drug: Levocetirizine ODT 5 mg
- Subjects of Group D: Part 2 (Experimental): Subjects in Group D will be randomized to receive levocetirizine ODT 5 mg without water in fasted state in Period 1. After a washout period of at least 5 days, subjects will receive levocetirizine IRT 5 mg with 150 mL water in fasted state in Period 2.
  Interventions: Drug: Levocetirizine IRT 5 mg; Drug: Levocetirizine ODT 5 mg

INTERVENTIONS:
Drug: Levocetirizine IRT 5 mg — Levocetirizine IRT will be available as film-coated tablets. Subjects will receive a single dose of 5 mg levocetirizine IRT. Subjects will receive levocetirizine IRT with 150 mL water in both Part (1 and 2).
Drug: Levocetirizine ODT 5 mg — Levocetirizine ODT will be available as oral disintegrating tablet. Subjects will receive a single dose of 5 mg levocetirizine ODT. In Part 1, subjects will receive levocetirizine ODT with 150 mL water and in Part 2 subjects will receive levocetirizine ODT without water.

SUMMARY:
This study will be an open-label, randomized 2-way cross-over study to evaluate bioequivalence study between levocetirizine ODT and levocetirizine IRT in healthy Japanese male subjects. Approximately 48 subjects will participate in this study to receive a single dose treatments of levocetirizine ODT 5 milligram (mg) or levocetirizine IRT 5 mg. In Part 1, subjects will randomized in 1:1 ratio (12 in each Period) in Period 1 and 2 to receive single dose of levocetirizine ODT 5 mg with water or single dose levocetirizine IRT 5 mg with water in fasted state. In this part, comparison of bioavailability of levocetirizine ODT and levocetirizine IRT when taken with water in the fasted state will be assessed. In Part 2, subjects will be randomized in 1:1 ratio (12 in each Period) in Period 1 and 2 to receive single dose levocetirizine ODT 5 mg without water or single dose levocetirizine IRT 5 mg with water in fasted state. In this part, comparison of bioavailability of levocetirizine ODT without water and levocetirizine IRT with water in the fasted state will be assessed. There will be at least a 5-day wash out period between the intervention periods. The duration of each subject's participation in each part will be approximately 7 weeks from screening to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 20 to 55 years of age inclusive, at the time of signing the informed consent.
* Japanese subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Subjects with body weight of >= 50 kilogram (kg) and body mass index (BMI) within the range of >=18.5 and <25.0 kg per meter square (m^2).
* In male subjects contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male subjects are eligible to participate if they agree to the following during the intervention period and until the completion of follow-ups: Refrain from donating sperm; Be abstinent from heterosexual or homosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; Agree to use a male condom and female partner to use an additional highly effective contraceptive method with a failure rate of <1 percentage per year when having sexual intercourse with a woman of childbearing potential who is not currently pregnant; Agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person.
* Subjects must be non-smokers.
* Subjects capable of giving signed informed consent.

Exclusion Criteria:

* Subjects with history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Subjects with abnormal blood pressure as determined by the investigator.
* Subjects with history of allergic rhinitis.
* Subjects with ALT >1.5x upper limit of normal (ULN).
* Subjects with bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percentage).
* Subjects with current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with QTc >450 millisecond (msec).
* Subjects with past or intended use of over-the-counter or prescription medication including vitamins, diet supplements (including St. John's wort), herbal medications within 14 days prior to first dosing or 5 half-lives (whichever is longer).
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation within 4 months prior to the first dosing day in this or any other clinical study involving an investigational study intervention or any other type of medical research (except for the subjects with no study intervention administered during any of those enrolment or participation).
* The subject with positive serological test for syphilis (Rapid Plasma Reagin [RPR] and Treponema pallidum [TP] antibody tests), Human immunodeficiency virus (HIV) Antigen/Antibody, Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody, or Human T-cell lymphotropic virus type 1 (HTLV-1) antibody at screening.
* Subject with positive pre-study drug screen.
* Subject with regular moderate alcohol consumption within 6 months prior to the study participation defined as: An average weekly intake of >14 units for males. One unit is equivalent to 360 milliliter (mL) of beer, 150 mL of wine or 45 mL of 80 proof distilled of spirits.
* Smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates participation in the study.
* History of donation of blood or blood products >= 400 mL within 3 months or >=200 mL within 1 month prior to the first dosing day.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Japanese male subjects will be part of this study.
Enrollment: 72 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single center, single dose, open-label, randomized, 2-part, 2-way crossover study. Bioequivalence (BE) between levocetirizine (levo) oral disintegrating tablet (ODT) and levocetirizine immediate release tablet (IRT) was evaluated in 72 healthy Japanese participants.
Pre-assignment Details: A total of 133 participants were screened, of them, 72 participants were randomized to receive study treatment. All participants except one participant randomized in Part 2 (Initial study) completed the study.
Groups:
- Part 1: Levo IRT 5 mg Followed by Levo ODT 5 mg (With Water): All participants received a single oral dose of levocetirizine IRT 5 milligram (mg) tablet with water in fasted state on Day 1 in Period 1. All participants received a single oral dose of levocetirizine ODT 5 mg tablet with water in fasted state on Day 1 in period 2. There was a washout period of at least 5 days between 2 periods.
- Part 1: Levo ODT 5 mg (With Water) Followed by Levo IRT 5 mg: All participants received a single oral dose of levocetirizine ODT 5 mg tablet with water in fasted state on Day 1 in Period 1. All participants received a single oral dose of levocetirizine IRT 5 mg tablet with water in fasted state on Day 1 in period 2. There was a washout period of at least 5 days between 2 periods.
- Part 2:Levo IRT 5 mg Followed by Levo ODT 5 mg (Without Water): All participants received a single oral dose of levocetirizine IRT 5 mg tablet with water in fasted state on Day 1 in Period 1. All participants received a single oral dose of levocetirizine ODT 5 mg tablet without water in fasted state on Day 1 in period 2. There was a washout period of at least 5 days between 2 periods.
- Part 2:Levo ODT 5 mg (Without Water) Followed by Levo IRT 5 mg: All participants received a single oral dose of levocetirizine ODT 5 mg tablet without water in fasted state on Day 1 in Period 1. All participants received a single oral dose of levocetirizine IRT 5 mg tablet with water in fasted state on Day 1 in period 2. There was a washout period of at least 5 days between 2 periods.
Period: Part 1:Treatment Period 1 (3 Days)
Arm/Group | Part 1: Levo IRT 5 mg Followed by Levo ODT 5 mg (With Water) | Part 1: Levo ODT 5 mg (With Water) Followed by Levo IRT 5 mg | Part 2:Levo IRT 5 mg Followed by Levo ODT 5 mg (Without Water) | Part 2:Levo ODT 5 mg (Without Water) Followed by Levo IRT 5 mg
Started | 12 | 12 | 0 | 0
Completed | 12 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1:Washout Period (at Least 5 Days)
Arm/Group | Part 1: Levo IRT 5 mg Followed by Levo ODT 5 mg (With Water) | Part 1: Levo ODT 5 mg (With Water) Followed by Levo IRT 5 mg | Part 2:Levo IRT 5 mg Followed by Levo ODT 5 mg (Without Water) | Part 2:Levo ODT 5 mg (Without Water) Followed by Levo IRT 5 mg
Started | 12 | 12 | 0 | 0
Completed | 12 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1:Treatment Period 2 (10 Days)
Arm/Group | Part 1: Levo IRT 5 mg Followed by Levo ODT 5 mg (With Water) | Part 1: Levo ODT 5 mg (With Water) Followed by Levo IRT 5 mg | Part 2:Levo IRT 5 mg Followed by Levo ODT 5 mg (Without Water) | Part 2:Levo ODT 5 mg (Without Water) Followed by Levo IRT 5 mg
Started | 12 | 12 | 0 | 0
Completed | 12 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2:Treatment Period 1 (3 Days)
Arm/Group | Part 1: Levo IRT 5 mg Followed by Levo ODT 5 mg (With Water) | Part 1: Levo ODT 5 mg (With Water) Followed by Levo IRT 5 mg | Part 2:Levo IRT 5 mg Followed by Levo ODT 5 mg (Without Water) | Part 2:Levo ODT 5 mg (Without Water) Followed by Levo IRT 5 mg
Started | 0 | 0 | 24 | 24
Completed | 0 | 0 | 24 | 24
Not Completed | 0 | 0 | 0 | 0
Period: Part 2:Washout Period (at Least 5 Days)
Arm/Group | Part 1: Levo IRT 5 mg Followed by Levo ODT 5 mg (With Water) | Part 1: Levo ODT 5 mg (With Water) Followed by Levo IRT 5 mg | Part 2:Levo IRT 5 mg Followed by Levo ODT 5 mg (Without Water) | Part 2:Levo ODT 5 mg (Without Water) Followed by Levo IRT 5 mg
Started | 0 | 0 | 24 | 24
Completed | 0 | 0 | 24 | 23
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Part 2:Treatment Period 2 (10 Days)
Arm/Group | Part 1: Levo IRT 5 mg Followed by Levo ODT 5 mg (With Water) | Part 1: Levo ODT 5 mg (With Water) Followed by Levo IRT 5 mg | Part 2:Levo IRT 5 mg Followed by Levo ODT 5 mg (Without Water) | Part 2:Levo ODT 5 mg (Without Water) Followed by Levo IRT 5 mg
Started | 0 | 0 | 24 | 23
Completed | 0 | 0 | 24 | 23
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Levo IRT 5 mg Followed by Levo ODT 5 mg (With Water) | Part 1: Levo ODT 5 mg (With Water) Followed by Levo IRT 5 mg | Part 2:Levo IRT 5 mg Followed by Levo ODT 5 mg (Without Water) | Part 2:Levo ODT 5 mg (Without Water) Followed by Levo IRT 5 mg | Total
Number analyzed (Participants) | 12 | 12 | 24 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.5 (6.72) | 31.8 (8.93) | 27.0 (7.00) | 26.3 (6.48) | 28.0 (7.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 12 | 12 | 24 | 24 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Japanese Heritage | 12 | 12 | 24 | 24 | 72

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Concentration-time Curve (AUC) From Time Zero Time (Pre-dose) to the Time of Last Quantifiable Concentration (AUC[0-t]) of Levocetirizine
Description: Blood samples were collected to measure AUC(0-t) at indicated time-points. AUC(0-t) was calculated by the linear trapezoidal method (i.e., Linear Trapezoidal Linear Interpolation calculation method in Phoenix WinNonlin).
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48 hours post-dose
Population: Pharmacokinetic (PK) Population is defined as all participants who were administered at least one dose of study treatment and blood samples for plasma drug concentration were taken and analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours*nanogram per milliliter (Hr*ng/mL)
Groups:
- Part 1: Levocetirizine ODT 5 mg: All participants received a single oral dose of levocetirizine ODT 5 mg tablet with water in fasted state either in Period 1 or Period 2 as per randomization schedule.
- Part 1: Levocetirizine IRT 5 mg: All participants received a single oral dose of levocetirizine IRT 5 mg tablet with water in fasted state either in Period 1 or Period 2 as per randomization schedule.
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Hours*nanogram per milliliter (Hr*ng/mL) | 1758.5 [1616.5 to 1913.0] | 1803.2 [1678.8 to 1936.8]
Statistical Analysis 1: Comparison: Part 1: Levocetirizine ODT 5 mg vs Part 1: Levocetirizine IRT 5 mg; Test type: Equivalence — If the 90 percent (%) confidence interval of the geometric mean ratio (Levocetirizine ODT/ Levocetirizine IRT) was within the acceptable range of 0.80 to 1.25 then Levocetirizine ODT was to be considered bioequivalent to the Levocetirizine IRT; Ratio of geometric mean = 0.975, 90% CI 2-sided [0.948 to 1.003]

2. Primary Outcome: Part 2: AUC(0-t) of Levocetirizine
Description: as for outcome 1
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hr*ng/mL
Groups:
- Part 2: Levocetirizine ODT 5 mg: All participants received a single oral dose of levocetirizine ODT 5 mg tablet without water in fasted state either in Period 1 or Period 2 as per randomization schedule.
- Part 2: Levocetirizine IRT 5 mg: All participants received a single oral dose of levocetirizine IRT 5 mg tablet with water in fasted state either in Period 1 or Period 2 as per randomization schedule.
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Hr*ng/mL | 1809.9 [1715.8 to 1909.2] | 1843.5 [1748.3 to 1943.9]
Statistical Analysis 1: Comparison: Part 2: Levocetirizine ODT 5 mg vs Part 2: Levocetirizine IRT 5 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric mean = 0.978, 90% CI 2-sided [0.958 to 0.998]

3. Primary Outcome: Part 1: Maximum Observed Concentration (Cmax) of Levocetirizine
Description: Blood samples were collected at indicated time points for analysis of Cmax. The values for Cmax were obtained directly from the concentration-time data.
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48 hours post-dose
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Nanogram per milliliter (ng/mL) | 219.9 [202.2 to 239.2] | 235.4 [214.2 to 258.7]
Statistical Analysis 1: Comparison: Part 1: Levocetirizine ODT 5 mg vs Part 1: Levocetirizine IRT 5 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric mean = 0.934, 90% CI 2-sided [0.875 to 0.998]

4. Primary Outcome: Part 2: Cmax of Levocetirizine
Description: as for outcome 3
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
ng/mL | 191.5 [181.8 to 201.8] | 223.6 [207.8 to 240.5]
Statistical Analysis 1: Comparison: Part 2: Levocetirizine ODT 5 mg vs Part 2: Levocetirizine IRT 5 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric mean = 0.857, 90% CI 2-sided [0.815 to 0.902]

5. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Zero Time (Pre-dose) Extrapolated to Infinite Time AUC(0-inf) of Levocetirizine
Description: Blood samples were collected at indicated time points for analysis of AUC(0-inf). AUC(0-inf)) of levocetirizine was calculated by standard non-compartmental analysis using the currently supported version of WinNonlin (version 6.3 or higher).
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Hr*ng/mL
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Hr*ng/mL | 1812.9 [1662.9 to 1976.3] | 1852.5 [1721.0 to 1994.0]

6. Secondary Outcome: Part 2: AUC(0-inf) of Levocetirizine
Description: Blood samples were collected at indicated time points for analysis of AUC(0-inf). AUC(0-inf) of levocetirizine was calculated by standard non-compartmental analysis using the currently supported version of WinNonlin (version 6.3 or higher).
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hr*ng/mL
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Hr*ng/mL | 1869.5 [1768.7 to 1976.0] | 1900.2 [1798.1 to 2008.2]

7. Secondary Outcome: Part 1: Time to First Occurrence of Cmax (Tmax) of Levocetirizine
Description: Blood samples were collected at indicated time points for analysis of tmax. The tmax of levocetirizine was obtained directly from the concentration-time data. The tmax was analyzed with the non-parametric Wilcoxon Matched Pairs Method (Signed Rank Method) to compute point estimate and associated 90% confidence interval for the median difference.
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Hours | 0.5000 [0.500 to 1.500] | 0.7500 [0.500 to 1.500]

8. Secondary Outcome: Part 2: Tmax of Levocetirizine
Description: as for outcome 7
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Hours | 1.0000 [0.500 to 4.000] | 1.0000 [0.500 to 3.000]

9. Secondary Outcome: Part 1: Apparent Terminal Phase Half-life (t1/2) of Levocetirizine
Description: Blood samples were collected at indicated time points for analysis of t1/2. The t1/2 of levocetirizine was calculated by standard non-compartmental analysis using the currently supported version of WinNonlin (version 6.3 or higher).
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Hours | 8.784 [8.143 to 9.475] | 8.544 [7.945 to 9.187]

10. Secondary Outcome: Part 2: t1/2 of Levocetirizine
Description: as for outcome 9
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Hours | 9.024 [8.611 to 9.458] | 8.933 [8.545 to 9.338]

11. Secondary Outcome: Part 1: Percentage of AUC(0-inf) Obtained by Extrapolation (%AUCex) of Levocetirizine
Description: Blood samples were collected at indicated time points for analysis of %AUCex. Percentage AUCex of levocetirizine was calculated by standard non-compartmental analysis using the currently supported version of WinNonlin (version 6.3 or higher).
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage AUCex
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Percentage AUCex | 2.772 [2.354 to 3.264] | 2.500 [2.156 to 2.898]

12. Secondary Outcome: Part 2: %AUCex of Levocetirizine
Description: as for outcome 11
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage AUCex
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Percentage AUCex | 2.973 [2.678 to 3.301] | 2.779 [2.501 to 3.089]

13. Secondary Outcome: Part 1: Apparent Clearance Following Oral Dosing (CL/F) of Levocetirizine
Description: Blood samples were collected at indicated time points for analysis of CL/F. CL/F of levocetirizine was calculated by standard non-compartmental analysis using the currently supported version of WinNonlin (version 6.3 or higher).
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Liters per hour
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Liters per hour | 2.758 [2.530 to 3.007] | 2.699 [2.507 to 2.905]

14. Secondary Outcome: Part 2: CL/F of Levocetirizine
Description: as for outcome 13
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Liters per hour
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Liters per hour | 2.675 [2.530 to 2.827] | 2.631 [2.490 to 2.781]

15. Secondary Outcome: Part 1: Apparent Volume of Distribution Following Oral Dosing (Vz/F) of Levocetirizine
Description: Blood samples were collected at indicated time points for analysis of Vz/F. Vz/F of levocetirizine was calculated by standard non-compartmental analysis using the currently supported version of WinNonlin (version 6.3 or higher).
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Liters | 34.95 [33.00 to 37.02] | 33.27 [31.55 to 35.08]

16. Secondary Outcome: Part 2: Vz/F of Levocetirizine
Description: Blood samples were collected at indicated time points for analysis of Vz/F. Vz/F of levocetirizine was calculated as by standard non-compartmental analysis using the currently supported version of WinNonlin (version 6.3 or higher).
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Liters | 34.82 [33.54 to 36.14] | 33.91 [32.60 to 35.27]

17. Secondary Outcome: Part 1: Elimination Rate Constant (Kel) (lambda_z) of Levocetirizine
Description: Blood samples were collected at indicated time points for analysis of kel. kel (lambda_z) is the first order rate constant associated with the terminal (log-linear) portion of the curve. kel of levocetirizine was calculated by standard non-compartmental analysis using the currently supported version of WinNonlin (version 6.3 or higher).
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Per hour
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Per hour | 0.07891 [0.07316 to 0.08512] | 0.08113 [0.07545 to 0.08724]

18. Secondary Outcome: Part 2: Kel (lambda_z) of Levocetirizine
Description: as for outcome 17
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Per hour
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Per hour | 0.07681 [0.07329 to 0.08050] | 0.07760 [0.07422 to 0.08112]

19. Secondary Outcome: Part 1: Mean Residence Time (MRT) of Levocetirizine
Description: Blood samples were collected at indicated time points for analysis of MRT. MRT of levocetirizine was calculated by standard non-compartmental analysis using the currently supported version of WinNonlin (version 6.3 or higher).
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Hours | 11.545 [10.649 to 12.516] | 11.417 [10.629 to 12.265]

20. Secondary Outcome: Part 2: MRT of Levocetirizine
Description: as for outcome 19
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Hours | 12.573 [11.991 to 13.182] | 12.272 [11.727 to 12.841]

21. Secondary Outcome: Part 1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is defined as any untoward medical occurrence that, at any dose may results in death or is life-threatening or requires inpatient hospitalization or results in persistent disability/incapacity or is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: Up to 18 days
Population: Safety Population consists of all participants who were administered at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Participants
  AEs | 0 | 0
  SAEs | 0 | 0

22. Secondary Outcome: Part 2: Number of Participants With AEs and SAEs
Description: as for outcome 21
Time Frame: Up to 18 days
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Participants
  AEs | 6 | 0
  SAEs | 0 | 0

23. Secondary Outcome: Part 1: Change From Baseline in Albumin and Total Protein Levels
Description: Blood samples were collected for the assessment of clinical chemistry parameters. Change from Baseline in albumin and total protein levels were evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Grams per liter (g/L)
  Albumin | 1.6 (1.64) | 1.5 (1.59)
  Total protein | 2.7 (2.16) | 2.3 (2.26)

24. Secondary Outcome: Part 2: Change From Baseline in Albumin and Total Protein Levels
Description: as for outcome 23
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
g/L
  Albumin | 1.2 (2.08) | 1.4 (2.17)
  Total protein | 1.8 (3.02) | 1.9 (3.34)

25. Secondary Outcome: Part 1: Change From Baseline in Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, Creatine Kinase, Gamma Glutamyl Transferase and Lactate Dehydrogenase Levels
Description: Blood samples were collected for the assessment of clinical chemistry parameters. Change from Baseline in alkaline phosphatase, alanine amino transferase, aspartate amino transferase, creatine kinase, gamma glutamyl transferase and lactate dehydrogenase levels were evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
International units per liter (IU/L)
  Alkaline phosphatase | -0.8 (8.08) | -1.6 (7.81)
  Alanine amino transferase | 0.5 (3.51) | 1.0 (3.32)
  Aspartate amino transferase | -0.1 (2.81) | -0.3 (2.05)
  Creatine kinase | -10.0 (29.62) | -13.2 (11.77)
  Gamma glutamyl transferase | -0.6 (1.06) | -0.5 (1.82)
  Lactate dehydrogenase | -11.0 (21.05) | -8.8 (10.10)

26. Secondary Outcome: Part 2: Change From Baseline in Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, Creatine Kinase, Gamma Glutamyl Transferase and Lactate Dehydrogenase Levels
Description: as for outcome 25
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
IU/L
  Alkaline phosphatase | -1.1 (13.46) | -2.3 (14.17)
  Alanine amino transferase | -0.5 (2.05) | -0.7 (2.63)
  Aspartate amino transferase | 0.1 (1.65) | -0.1 (2.58)
  Creatine kinase | -12.4 (16.24) | -16.3 (20.93)
  Gamma glutamyl transferase | -0.1 (1.28) | -0.1 (1.52)
  Lactate dehydrogenase | -3.5 (10.52) | -3.7 (11.55)

27. Secondary Outcome: Part 1: Change From Baseline in Amylase Levels
Description: Blood samples were collected for the assessment of clinical chemistry parameters. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Units per liter (U/L) | 6.3 (7.94) | 7.2 (10.62)

28. Secondary Outcome: Part 2: Change From Baseline in Amylase Levels
Description: Blood samples were collected for the assessment of clinical chemistry parameters. Change from Baseline in amylase levels were evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
U/L | 7.4 (6.69) | 7.1 (10.13)

29. Secondary Outcome: Part 1: Change From Baseline in Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid Levels
Description: Blood samples were collected for the assessment of clinical chemistry parameters. Change from Baseline in direct bilirubin, total bilirubin, creatinine and uric acid levels were evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter (UMOL/L)
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Micromoles per liter (UMOL/L)
  Direct bilirubin | 0.214 (0.9178) | 0.356 (1.0059)
  Total bilirubin | 0.143 (3.3034) | -1.710 (4.0340)
  Creatinine | -1.9522 (4.20313) | -1.9890 (4.09064)
  Uric acid | 21.0658 (22.25394) | 23.2963 (27.33699)

30. Secondary Outcome: Part 2: Change From Baseline in Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid Levels
Description: as for outcome 29
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: UMOL/L
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
UMOL/L
  Direct bilirubin | -0.071 (0.7018) | 0.036 (0.7555)
  Total bilirubin | -0.748 (3.0325) | -0.619 (3.1374)
  Creatinine | -3.5913 (4.21949) | -3.8746 (5.00254)
  Uric acid | 14.0026 (20.14225) | 13.6677 (28.30678)

31. Secondary Outcome: Part 1: Change From Baseline in Calcium, Cholesterol, Chloride, Glucose, High Density Lipids Cholesterol, Potassium, Low Density Lipids Cholesterol, Sodium, Phosphorus Inorganic, Triglycerides and Urea/Blood Urea Nitrogen (BUN) Levels
Description: Blood samples were collected for the assessment of clinical chemistry parameters. Change from Baseline in calcium, cholesterol, chloride, glucose, high density lipids cholesterol, potassium, low density lipids cholesterol, sodium, phosphorus inorganic, triglycerides and urea/blood urea nitrogen (BUN) levels were evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (MMOL/L)
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Millimoles per liter (MMOL/L)
  Calcium | 0.032227 (0.0490682) | 0.018713 (0.0594308)
  Cholesterol | 0.117448 (0.2967150) | 0.054953 (0.2589722)
  Chloride | -0.9 (1.19) | -1.0 (1.43)
  Glucose | -0.067075 (0.2724243) | -0.050884 (0.2037377)
  High density lipids cholesterol | -0.032325 (0.1006621) | -0.063573 (0.0806953)
  Potassium | 0.13 (0.311) | 0.10 (0.330)
  Low density lipids cholesterol | 0.059263 (0.2661881) | 0.038790 (0.2158221)
  Sodium | -0.6 (1.24) | -0.7 (1.49)
  Phosphorus inorganic | -0.193740 (0.0737556) | -0.182977 (0.0849880)
  Triglycerides | 0.04520 (0.284839) | -0.00047 (0.304261)
  Urea/BUN | 0.01934 (0.472088) | 0.08033 (0.498940)

32. Secondary Outcome: Part 2: Change From Baseline in Calcium, Cholesterol, Chloride, Glucose, High Density Lipids Cholesterol, Potassium, Low Density Lipids Cholesterol, Sodium, Phosphorus Inorganic, Triglycerides and Urea/BUN Levels
Description: Blood samples were collected for the assessment of clinical chemistry parameters. Change from Baseline in calcium, cholesterol, chloride, glucose, high density lipids cholesterol, potassium, low density lipids cholesterol, sodium, phosphorus inorganic, triglycerides and urea/BUN levels were evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: MMOL/L
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
MMOL/L
  Calcium | 0.015594 (0.0623219) | 0.015926 (0.0704590)
  Cholesterol | 0.083506 (0.2666316) | 0.064925 (0.2594347)
  Chloride | -0.6 (1.17) | -0.5 (1.35)
  Glucose | -0.049728 (0.2525006) | 0.059053 (0.2990211)
  High density lipids cholesterol | -0.049565 (0.1151357) | -0.047869 (0.0975044)
  Potassium | -0.03 (0.233) | 0.08 (0.368)
  Low density lipids cholesterol | 0.123374 (0.1986158) | 0.084733 (0.1846539)
  Sodium | -1.1 (1.28) | -0.6 (1.05)
  Phosphorus inorganic | -0.203831 (0.1251750) | -0.239770 (0.1230018)
  Triglycerides | -0.02707 (0.290907) | 0.03606 (0.206604)
  Urea/BUN | -0.12272 (0.622969) | -0.45802 (0.817628)

33. Secondary Outcome: Part 1: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes and Total Neutrophils Count
Description: Blood samples were collected for the assessment of hematology parameters. Change from Baseline in basophils, eosinophils, lymphocytes, monocytes and total neutrophils levels were evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Percentage
  Basophils | -0.01 (0.150) | 0.01 (0.212)
  Eosinophils | -0.53 (0.783) | -0.52 (1.087)
  Lymphocytes | -5.94 (6.330) | -5.96 (7.705)
  Monocytes | -0.16 (0.835) | 0.16 (1.443)
  Total neutrophils levels | 6.64 (6.480) | 6.32 (7.950)

34. Secondary Outcome: Part 2: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes and Total Neutrophils Count
Description: as for outcome 33
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Percentage
  Basophils | 0.08 (0.195) | 0.04 (0.176)
  Eosinophils | -0.92 (1.183) | -0.74 (1.012)
  Lymphocytes | -8.45 (6.915) | -8.07 (5.558)
  Monocytes | -0.49 (1.046) | -0.48 (1.087)
  Total neutrophils levels | 9.78 (7.094) | 9.25 (5.847)

35. Secondary Outcome: Part 1: Change From Baseline in Platelet Count and White Blood Cell Count
Description: Blood samples were collected for the assessment of hematology parameters. Change from Baseline in platelet count and white blood cell count were evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Giga per liter (GI/L)
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Giga per liter (GI/L)
  Platelet count | -6.4 (12.62) | -11.4 (11.64)
  White blood cell count | -0.94 (0.950) | -1.26 (0.596)

36. Secondary Outcome: Part 2: Change From Baseline in Platelet Count and White Blood Cell Count
Description: as for outcome 35
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
GI/L
  Platelet count | -2.5 (12.71) | -2.9 (13.98)
  White blood cell count | -1.14 (1.246) | -1.06 (1.133)

37. Secondary Outcome: Part 1: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration
Description: Blood samples were collected for the assessment of hematology parameters. Change from Baseline in hemoglobin and mean corpuscle hemoglobin concentration were evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Grams per liter (G/L)
  Hemoglobin | 2.2 (3.81) | 2.3 (3.44)
  Mean corpuscle hemoglobin concentration | 2.3 (4.16) | 1.8 (4.64)

38. Secondary Outcome: Part 2: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration
Description: as for outcome 37
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
G/L
  Hemoglobin | 0.9 (4.87) | 0.9 (5.69)
  Mean corpuscle hemoglobin concentration | 0.2 (4.12) | 0.5 (3.87)

39. Secondary Outcome: Part 1: Change Form Baseline in Hematocrit
Description: Blood samples were collected for the assessment of hematology parameters. Change from Baseline in hematocrit was evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Proportion of red blood cells in blood | 0.0036 (0.01014) | 0.0043 (0.00952)

40. Secondary Outcome: Part 2: Change Form Baseline in Hematocrit
Description: as for outcome 39
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Proportion of red blood cells in blood | 0.0023 (0.01505) | 0.0019 (0.01595)

41. Secondary Outcome: Part 1: Change From Baseline in Mean Corpuscle Hemoglobin
Description: Blood samples were collected for the assessment of hematology parameters. Change from Baseline in mean corpuscle hemoglobin was evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Picograms | -0.04 (0.313) | -0.03 (0.288)

42. Secondary Outcome: Part 2: Change From Baseline in Mean Corpuscle Hemoglobin
Description: as for outcome 41
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Picograms | -0.07 (0.305) | -0.07 (0.265)

43. Secondary Outcome: Part 1: Change From Baseline in Mean Corpuscle Volume
Description: Blood samples were collected for the assessment of hematology parameters. Change from Baseline in mean corpuscle volume was evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Femtoliters | -0.6 (0.83) | -0.5 (0.83)

44. Secondary Outcome: Part 2: Change From Baseline in Mean Corpuscle Volume
Description: as for outcome 43
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Femtoliters | -0.2 (0.81) | -0.3 (0.63)

45. Secondary Outcome: Part 1: Change From Baseline in Red Blood Cell Count
Description: Blood samples were collected for the assessment of hematology parameters. Change from Baseline in red blood cell count was evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Trillion cells per liter | 0.078 (0.1189) | 0.080 (0.1235)

46. Secondary Outcome: Part 2: Change From Baseline in Red Blood Cell Count
Description: as for outcome 45
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Trillion cells per liter | 0.040 (0.1730) | 0.041 (0.1883)

47. Secondary Outcome: Part 1: Change From Baseline in Reticulocytes
Description: Blood samples were collected for the assessment of hematology parameters. Change from Baseline in reticulocytes was evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Percentage of reticulocytes | -0.0001 (0.00167) | 0.0004 (0.00186)

48. Secondary Outcome: Part 2: Change From Baseline in Reticulocytes
Description: as for outcome 47
Time Frame: Baseline (Day 1, Pre-dose) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Percentage of reticulocytes | -0.0001 (0.00173) | -0.0004 (0.00169)

49. Secondary Outcome: Part 1: Number of Participants With Urinalysis Results by Dipstick Method
Description: Urine samples were collected to assess urine bilirubin, urine occult blood, urine glucose, urine ketones, urine protein and urine urobilinogen by dipstick test. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameter of urine bilirubin, urine occult blood, urine glucose, urine ketones, urine protein and urine urobilinogen can be read as negative (-), trace and 1+ indicating proportional concentrations in the urine sample. Only categories with significant values have been presented.
Time Frame: Pre-dose (Day 1) and 48 hours post-dose
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Participants
  Bilirubin, Pre-dose, negative | 24 | 24
  Bilirubin, 48 hours, negative | 24 | 24
  Occult blood, Pre-dose, negative | 23 | 24
  Occult blood, Pre-dose, trace | 1 | 0
  Occult blood, 48 hours, negative | 23 | 24
  Occult blood, 48 hours, trace | 1 | 0
  Glucose, Pre-dose, negative | 24 | 24
  Glucose, 48 hours, negative | 24 | 24
  Ketones, Pre-dose, negative | 24 | 23
  Ketones, Pre-dose, positive (1+) | 0 | 1
  Ketones, 48 hours, negative | 24 | 24
  Protein, Pre-dose, negative | 24 | 24
  Protein, 48 hours, negative | 24 | 24
  Urobilinogen, Pre-dose, trace | 24 | 24
  Urobilinogen, 48 hours, trace | 24 | 24

50. Secondary Outcome: Part 2: Number of Participants With Urinalysis Results by Dipstick Method
Description: as for outcome 49
Time Frame: Pre-dose (Day 1) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Participants
  Bilirubin, Pre-dose, negative | 48 | 47
  Bilirubin, 48 hours, negative | 48 | 47
  Occult blood, Pre-dose, negative | 48 | 47
  Occult blood, 48 hours, negative | 47 | 47
  Occult blood, 48 hours, trace | 1 | 0
  Glucose, Pre-dose, negative | 48 | 47
  Glucose, 48 hours, negative | 48 | 47
  Ketones, Pre-dose, negative | 48 | 46
  Ketones, Pre-dose, positive (1+) | 0 | 1
  Ketones, 48 hours, negative | 48 | 47
  Protein, Pre-dose, negative | 48 | 47
  Protein, 48 hours, negative | 48 | 47
  Urobilinogen, Pre-dose, trace | 48 | 47
  Urobilinogen, 48 hours, trace | 48 | 47

51. Secondary Outcome: Part 1: Urine Potential of Hydrogen (pH)
Description: Urine samples were collected for the measurement of urine pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0).
Time Frame: Pre-dose (Day 1) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
pH
  Pre-dose | 6.04 (0.359) | 6.06 (0.340)
  48 hours | 6.10 (0.329) | 6.02 (0.275)

52. Secondary Outcome: Part 2: Urine Potential of Hydrogen (pH)
Description: as for outcome 51
Time Frame: Pre-dose (Day 1) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
pH
  Pre-dose | 6.20 (0.353) | 6.11 (0.345)
  48 hours | 6.09 (0.395) | 6.00 (0.376)

53. Secondary Outcome: Part 1: Urine Specific Gravity
Description: Urine samples were collected for the measurement of specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. The urinary specific gravity measurement is a routine part of urinalysis. The reference range is 1.002-1.030.
Time Frame: Pre-dose (Day 1) and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Ratio
  Pre-dose | 1.0158 (0.00724) | 1.0144 (0.00658)
  48 hours | 1.0178 (0.00751) | 1.0163 (0.00798)

54. Secondary Outcome: Part 2: Urine Specific Gravity
Description: as for outcome 53
Time Frame: Pre-dose (Day 1) and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Ratio
  Pre-dose | 1.0156 (0.00646) | 1.0179 (0.00666)
  48 hours | 1.0160 (0.00669) | 1.0159 (0.00749)

55. Secondary Outcome: Part 1: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured in supine position after 5 minutes rest. Change from Baseline in SBP and DBP was evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 1, 24, 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Millimeters of mercury (mmHg)
  SBP, 1 hour | -2.0 (9.68) | 0.4 (8.54)
  SBP, 24 hour | 0.0 (7.23) | 0.6 (7.20)
  SBP, 48 hour | -1.2 (9.64) | 1.3 (7.51)
  DBP, 1 hour | -1.8 (5.67) | -2.2 (6.84)
  DBP, 24 hour | 0.3 (4.47) | 0.0 (6.19)
  DBP, 48 hour | 0.6 (6.98) | 1.1 (6.10)

56. Secondary Outcome: Part 2: Change From Baseline in SBP and DBP
Description: as for outcome 55
Time Frame: Baseline (Day 1, Pre-dose) and 1, 24, 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
mmHg
  SBP, 1 hour | 0.2 (9.22) | -0.9 (8.27)
  SBP, 24 hour | -1.9 (7.69) | -1.2 (9.16)
  SBP, 48 hour | 0.7 (9.95) | 0.3 (9.15)
  DBP, 1 hour | -2.6 (7.07) | -2.6 (6.35)
  DBP, 24 hour | -2.3 (6.11) | -1.2 (6.23)
  DBP, 48 hour | -0.6 (7.15) | -0.2 (6.22)

57. Secondary Outcome: Part 1: Change From Baseline in Heart Rate
Description: Heart rate was measured in supine position after 5 minutes rest. Change from Baseline in heart rate was evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 1, 24, 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Beats per minute
  1 hour | -2.3 (4.77) | -0.9 (4.62)
  24 hour | -0.8 (5.24) | -0.1 (5.50)
  48 hour | 0.8 (6.13) | 2.5 (5.90)

58. Secondary Outcome: Part 2: Change From Baseline in Heart Rate
Description: as for outcome 57
Time Frame: Baseline (Day 1, Pre-dose) and 1, 24, 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Beats per minute
  1 hour | -1.5 (8.34) | -0.6 (5.24)
  24 hour | -1.9 (9.16) | 0.6 (6.91)
  48 hour | 1.5 (10.85) | 3.0 (9.08)

59. Secondary Outcome: Part 1: Change From Baseline in Body Temperature
Description: Body temperature was measured in supine position after 5 minutes rest. Change from Baseline in body temperature was evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 1, 24, 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Degree Celsius
  1 hour | 0.20 (0.313) | 0.02 (0.392)
  24 hour | -0.01 (0.292) | 0.09 (0.268)
  48 hour | 0.06 (0.280) | 0.01 (0.307)

60. Secondary Outcome: Part 2: Change From Baseline in Body Temperature
Description: as for outcome 59
Time Frame: Baseline (Day 1, Pre-dose) and 1, 24, 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Degree Celsius
  1 hour | 0.19 (0.362) | 0.09 (0.359)
  24 hour | 0.13 (0.272) | 0.08 (0.324)
  48 hour | 0.03 (0.351) | 0.03 (0.345)

61. Secondary Outcome: Part 1: Change From Baseline in Heart Rate (12-Lead Electrocardiogram [ECG])
Description: Single 12-lead ECG was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT interval with Fridericia's correction (QTcF). Change from Baseline in heart rate (ECG) was evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 1, 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Beats per minute
  1 hour | 1.6 (4.80) | 1.0 (4.47)
  48 hour | 2.1 (4.37) | 2.5 (4.74)

62. Secondary Outcome: Part 2: Change From Baseline in Heart Rate (ECG)
Description: Single 12-lead ECG was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF. Change from Baseline in heart rate (ECG) was evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 1, 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Beats per minute
  1 hour | -1.0 (5.72) | -1.7 (5.83)
  48 hour | 1.7 (8.22) | 1.9 (8.05)

63. Secondary Outcome: Part 1: Change From Baseline in PR Interval, QRS Interval, QT Interval and QTcF Interval
Description: Single 12-lead ECG was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF. Change from Baseline in PR interval, QRS interval, QT interval and QTcF interval was evaluated. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and 1, 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 24 | 24
Millisecond
  PR interval, 1 hour | -7.3 (12.16) | -6.3 (10.00)
  PR interval, 48 hour | -5.5 (10.72) | -1.9 (13.03)
  QRS duration, 1 hour | -0.5 (3.40) | -0.8 (5.24)
  QRS duration, 48 hour | 1.7 (3.67) | -0.6 (6.37)
  QT interval, 1 hour | -9.3 (17.30) | -6.4 (15.38)
  QT interval, 48 hour | -14.3 (16.00) | -10.7 (18.17)
  QTcF interval, 1 hour | -6.1 (14.06) | -4.3 (11.52)
  QTcF interval, 48 hour | -9.3 (14.67) | -4.8 (17.96)

64. Secondary Outcome: Part 2: Change From Baseline in PR Interval, QRS Interval, QT Interval and QTcF Interval
Description: Single 12-lead ECG was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF. Change from Baseline in PR interval, QRS interval, QT interval and QTcF interval was evaluated. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. The Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and 1, 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
Number analyzed (Participants) | 48 | 47
Millisecond
  PR interval, 1 hour | -3.2 (11.67) | -2.8 (8.66)
  PR interval, 48 hour | 1.2 (11.48) | 0.6 (9.76)
  QRS duration, 1 hour | -1.4 (5.53) | -1.9 (7.99)
  QRS duration, 48 hour | 0.3 (6.50) | -0.4 (7.17)
  QT interval, 1 hour | 3.8 (14.45) | 3.1 (18.94)
  QT interval, 48 hour | -12.1 (17.36) | -11.4 (20.49)
  QTcF interval, 1 hour | 1.4 (15.35) | -0.9 (17.35)
  QTcF interval, 48 hour | -8.5 (15.75) | -7.6 (14.87)

ADVERSE EVENTS:
Time Frame: On-therapy non-SAEs and SAEs were reported from start of study treatment and up to 18 days
Description: Non-SAE and SAEs were reported for Safety Population. Adverse events were presented treatment-wise.
Arm/Group | Part 1: Levocetirizine ODT 5 mg | Part 1: Levocetirizine IRT 5 mg | Part 2: Levocetirizine ODT 5 mg | Part 2: Levocetirizine IRT 5 mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 6/48 | 0/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Levocetirizine ODT 5 mg (N=24) | Part 1: Levocetirizine IRT 5 mg (N=24) | Part 2: Levocetirizine ODT 5 mg (N=48) | Part 2: Levocetirizine IRT 5 mg (N=48)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT03555890/SAP_000.pdf
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03555890/Prot_001.pdf